CLINICAL TRIAL: NCT02178371
Title: Effects of Modified Constraint Induced Movement Therapy on Infantile Hemiplegia
Brief Title: Constraint Induced Movement Therapy on Infantile Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-006
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Hemiplegia
Keywords: Upper extremity; Physical therapy modalities
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UTWC (control group) (Experimental): the control group performs the same tasks than the experimental group, but without healthy hand constraint/containment.
  Interventions: Procedure: Unimanual therapy without constraint UTWC
- mCIMT (Experimental): The study is conducted over a period of 5 weeks of treatment, using a movement restriction time healthy upper extremity of 2 hours daily.
  The restriction applied in the study is performed with the closed hand position and thumb inside the fist through a transparent film that reaches the wrist joint.
  In periods mCIMT, monitored the activities designed to enhance their functionality, based on motivation, avoiding frustrations are made.
  Interventions: Procedure: mCIMT

INTERVENTIONS:
Procedure: mCIMT — affected upper limb use with constraint of the healthy hand
  Other Names: Modified constraint-induced movement therapy
  Arms: mCIMT
Procedure: Unimanual therapy without constraint UTWC — affected upper limb use without constraint of healthy hand
  Arms: UTWC (control group)

SUMMARY:
The purpose of this study is to assess the functionality of the affected upper limb in infantile hemiplegia by applying a protocol of modified constraint-induced movement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children's Hemiplegia Medical diagnosis.
* Aged between 4 and 8 years.
* Lack of activity of the affected upper extremity.
* Overcoming 10th extension at the metacarpophalangeal and interphalangeal joint.
* Complete the 20 º of wrist extension of the affected upper extremity.
* Adequate cognitive development to understand verbal commands given for the execution of tasks.
* Cooperation in the execution of tasks.

Exclusion Criteria:

* To Have vision problems that prevent them from carrying out the intervention.
* Having significant balance changes that endanger the child fall to bring a restriction in the affected upper limb.
* Submit uncontrolled seizures.
* To Have received botulinum toxin prior to 6 months prior to the intervention.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Quality of Upper Extremity Skills Test (QUEST) at week 5. | Baseline, week 5.
Change from baseline on the Shuee Evaluation at week 5 | baseline, week 5

SECONDARY OUTCOMES:
Change from baseline on visual-motor coordination at week 5. | Baseline, week 5.
  Circuit described by Mak in 2010
Change from baseline on Grip strength at week 5. | Baseline, week 5.
Change from baseline on the Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) at week 5. | Baseline, week 5.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Palomo Carrión, PhD, PT, Principal Investigator — San Pablo CEU University; Francisco García-Muro SAn José, PhD, PT, Study Director — San Pablo CEU University
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain